CLINICAL TRIAL: NCT03085849
Title: A Phase I Study Evaluating the Safety and Efficacy of SGI-110 Followed by Combined Durvalumab Plus Tremelimumab in Subjects With Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: SGI-110 Plus Durvalumab/Tremelimumab in SCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Shu (Other)
Responsible Party: Sponsor-Investigator, Catherine Shu, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ8257
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; tremelimumab; guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects with ES-SCLC, progressive after platinum-based first-line chemotherapy will receive SGI-110 followed by combined durvalumab plus tremelimumab.
  1. Dose escalation phase: 6-12 patients
  2. MTD expansion cohort: 10 patients
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: SGI-110

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV on day 8 (flat dose) until progression
  Other Names: MEDI4736
Drug: Tremelimumab — 75 mg IV on day 8 (flat dose) x 4 doses
  Other Names: CP-675,206
Drug: SGI-110 — SC daily for 5 days (days 1-5) until progression or toxicity
  Dose escalation scheme:
  Dose level -1 - SGI-110 20 mg/m2 SC daily; Dose level 0 - SGI-110 30 mg/m2 SC daily; Dose level 1 - SGI-110 45 mg/m2 SC daily; and SGI-110 given on days 1-5 of every 28 day cycle
  Other Names: Guadecitabine

SUMMARY:
The purpose of this study is to determine if a combination of investigational agents is safe to give to people with small cell lung cancer (SCLC) after standard chemotherapy has been attempted. Subjects enrolled in this trial will receive 3 investigational drugs: SGI-110 (guadecitabine), durvalumab (MEDI4736) and tremelimumab.

DETAILED DESCRIPTION:
SCLC accounts for approximately 15% of new cases of lung cancer, and an estimated 33,000 cases are expected to be diagnosed in the United States in 2016. Compared to NSCLC, SCLC typically has a more rapid doubling time, a higher growth fraction, and earlier development of distant metastases. Patients with limited stage (LS) disease are treated with curative intent using definitive, concurrent chemotherapy and thoracic radiotherapy. For patients with extensive stage (ES) disease, systemic chemotherapy can prolong survival in most cases, however long-term survival is rare. Despite the activity of several agents in SCLC, an etoposide plus platinum (i.e. cisplatin) doublet regimen remains the standard of care in the first-line setting because of its higher activity compared to other chemotherapy regimens, as well as the ease of combining it with radiation. Initial response rates may be as high as 70-90% in LS-SCLC and 50-70% in ES-SCLC. However, the disease typically recurs rapidly which is reflected by median survival rates of 9 to 11 months for ES-SCLC and a 2-year survival rate of less than 5%.

This study has a 3 + 3 design that will be used to assess the safety of SGI-110 given prior to flat doses of durvalumab (1500 mg) and tremelimumab (75 mg). The starting dose of SGI-110 will be 30 mg/m2 (dose level 0) and the target dose that is predicted to be safe and most effective will be 45 mg/m2 (dose level 1). These doses have been chosen based on safety and efficacy data from phase 1 clinical trials in other solid tumors, as described above. Patients enrolled in any given dose level will be evaluated for safety (adverse events monitoring) and efficacy. There will be mandatory pre- and on-treatment tumor biopsies performed in alternating fashion on cycle 1 day 8 +/- 2 days or cycle 2 day 8 +/- 2 days. The dose-limiting toxicity (DLT) observation period will last for 4 weeks (28 days) and ends on C2D1. Delayed serious immune-mediated adverse events will also be monitored but will not be considered dose limiting toxicities.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Written informed consent and any locally-required authorization (e.g., HIPAA in the USA, EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age ≥ 18 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG performance status of 0 or 1)
4. Life expectancy of ≥ 12 weeks
5. Adequate normal organ and marrow function as defined below Hemoglobin ≥ 9.0 g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3) Platelet count ≥ 100 x 109/L (>100,000 per mm3) Serum total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (for patients with a diagnosis of Gilbert's syndrome, direct bilirubin ≤ 1.5 x ULN) AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN

   Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) . 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
6. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 180 days after the final dose of investigational product. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Female subjects must also refrain from egg cell donation for 180 days after the final dose of investigational product.

   A) Females of childbearing potential are defined as those who are not surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are not postmenopausal (defined as 12 months with no menses with postmenopausal gonadotropin levels [luteinizing hormone and follicle-stimulating hormone], or estradiol levels within the postmenopausal range according to local guidelines without an alternative medical cause).

   B) A highly effective method of contraception is defined as one that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly.
7. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
8. Subjects must have a histologically confirmed diagnosis of small cell lung carcinoma. A fresh, pre-treatment tumor biopsy will be required to evaluate tumor infiltrating lymphocytes, PD-L1 IHC staining, methylation status, etc. as outlined in the study timeline. All subjects are also required to have a C1D8 (or C2D8) biopsy.
9. Subjects must have extensive-stage disease (by NCCN criteria) that is progressive or relapsed after platinum-based chemotherapy.
10. Tumor burden must be radiographically measurable by RECIST criteria.
11. At time of Day 1 of the study, subjects with central nervous system metastases must have been treated and must be asymptomatic and meet the following:

    1. No concurrent treatment, inclusive of but not limited to surgery, radiation, and/or corticosteroids
    2. Neurologic stability (lack of signs and symptoms greater than baseline prior to XRT) until the time of dosing
    3. For radiation treatment, there should be at least 14 days between the last day of stereotactic radiosurgery or gamma-knife treatment and Day 1 of protocol treatment. For WBRT, there should be at least 28 days between last day of WBRT and Day 1 of protocol treatment.
    4. Note: patients with leptomeningeal disease or cord compression are excluded from the study.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous enrollment in the present study.
3. Participation in another clinical study with an investigational product during the last 4 weeks.
4. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab or an anti-CTLA4, including tremelimumab
5. Any previous treatment with a hypomethylating agent, including decitabine, azacitidine, or SGI-110.
6. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study drug and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
7. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, gamma-knife, other investigational agent) ≤ 14 days prior to the first dose of study drug. For WBRT, the washout period is 28 days. Local treatment of isolated lesions for palliative RT (by radiotherapy, for example) is acceptable.
8. Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from electrocardiogram (in triplicate, if applicable) using Fredericia's Correction
9. Liver cirrhosis or chronic liver disease Childs-Pugh B or C.
10. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
11. Receipt of the tyrosine kinase inhibitor sunitinib within 90 days before the first dose of study therapy.
12. Any unresolved toxicity ( > CTCAE grade 2) from previous anti-cancer therapy.
13. Any prior Grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
14. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
15. Active or prior documented history of pneumonitis or interstitial lung disease.
16. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
17. History of primary immunodeficiency
18. History of allogeneic organ transplant
19. History of hypersensitivity to durvalumab, tremelimumab, SGI-110, or any excipient.
20. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
21. Known history of active tuberculosis
22. Leptomeningeal carcinomatosis or cord compression
23. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab
24. Female subjects who are pregnant or breast-feeding, or male or female patients of reproductive potential who are not willing to employ a highly effective method of contraception from screening to 180 days after the last dose of investigational therapy.
25. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
26. Symptomatic or uncontrolled brain metastases requiring concurrent treatment (surgery, RT, corticosteroids)
27. Subjects with uncontrolled seizures.
28. Concomitant use of drugs with laxative properties and/or herbal/natural remedies for constipation. These agents should be avoided for 90 days after the last dose of investigational therapy, given the potential for exacerbation of diarrhea.
29. Known significant mental illness or other conditions such as active alcohol or other substance abuse/addiction that, in the opinion of the investigator, predisposes the subject to high risk of noncompliance with the protocol.

Procedures for withdrawal of incorrectly enrolled patients are presented in Section 5.5.1. If a patient withdraws from participation in the study, then his or her enrollment/randomization code cannot be reused. Withdrawn patients will not be replaced.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of SGI-110 | Approximately 24 to 48 weeks
  Defined as the highest dose cohort for SGI-110 with a rate of dose limiting toxicity (DLT) <33%.

SECONDARY OUTCOMES:
Rate of treatment related adverse events | Up to 90 days after last study dose
  Defined by the percentage of patients receiving study treatment and experiencing grade 3-4 treatment related adverse events.
Overall Response Rate (ORR) | Up to 12 months after last study dose
  Defined by the proportion of patients with tumor size reduction of a predefined amount and for a minimum time period.
Median Progression Free Survival (mPFS) | Up to 24 months after last study dose
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. Estimated using the Kaplan-Meier method in number of weeks.
Median Overall Survival (mOS) | Up to 24 months after last study dose
  The length of time from the start of treatment for a disease, such as cancer, that half of the patients in a group of patients diagnosed with the disease are still alive. Estimated using the Kaplan-Meier method in number of weeks.
Median Duration of Response (mDOR) | Up to 12 months after last study dose
  Duration of overall response is measured from the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Shu, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Chute JP, Chen T, Feigal E, Simon R, Johnson BE. Twenty years of phase III trials for patients with extensive-stage small-cell lung cancer: perceptible progress. J Clin Oncol. 1999 Jun;17(6):1794-801. doi: 10.1200/JCO.1999.17.6.1794. PMID 10561217
- [Background] Janne PA, Freidlin B, Saxman S, Johnson DH, Livingston RB, Shepherd FA, Johnson BE. Twenty-five years of clinical research for patients with limited-stage small cell lung carcinoma in North America. Cancer. 2002 Oct 1;95(7):1528-38. doi: 10.1002/cncr.10841. PMID 12237922